CLINICAL TRIAL: NCT05268380
Title: Collision of Three Global Pandemics: the Effect of Tuberculosis and HIV on the Epidemiological, Clinical, Virological and Immunological Trajectory of COVID-19 in Botswana and Namibia
Acronym: Core-NB
Status: Completed | Type: Observational
Sponsor: University of Namibia (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Research Center Borstel (Other); Victus Global Botswana Organization (Unknown)
Responsible Party: Principal Investigator, Mareli Claassens, Associate research professor, University of Namibia
Other Study IDs: RIA2020EF-2963
Record Dates: First submitted 2022-03-02; First posted 2022-03-07 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; HIV Seropositivity; Tuberculosis, Pulmonary; Tuberculosis Infection
MeSH Terms: conditions — COVID-19; HIV Seropositivity; Tuberculosis, Pulmonary; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sputum, blood and nasopharyngeal swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Household contact study: Investigation of Covid-19 index cases' households for TB infection and disease, HIV seropositivity, Covid-19 active infection and previous infection.
  Interventions: Diagnostic Test: Covid-19, TB and HIV diagnosis
- Primary healthcare facility study: Investigation of primary healthcare facility attendees for TB infection and disease, HIV seropositivity, Covid-19 active infection and previous infection.
  Interventions: Diagnostic Test: Covid-19, TB and HIV diagnosis

INTERVENTIONS:
Diagnostic Test: Covid-19, TB and HIV diagnosis — GeneXpert (sputum) will be used to diagnose active TB disease, IGRA will be used to diagnose latent TB infection, PCR will be used to diagnose Covid-19 active infection, HIV rapid test will be used to diagnose HIV seropositivity.

SUMMARY:
COVID-19 has emerged as global pandemic during the past few months, with an unprecedented impact on public health, and society more generally. Virus epidemiology is poorly understood, as are factors influencing the diverse clinical picture. To date most cases have been seen in high income countries and consequently COVID-19 diagnostics and research have mainly been set-up in these settings. Outstanding questions include an understanding of how the virus spreads and how it causes pathology. A particular gap in current knowledge is the effect of HIV and tuberculosis (TB) on the outcomes of COVID-19 disease as these two conditions impair the host immune response to other infectious disease. Understanding how these three pandemics interact is crucial. We have developed a proposal that will answer critical questions concerning COVID-19 disease epidemiology in the context of low resource countries with high burden of poverty, and in the presence of high rates of TB and HIV, namely, Namibia and Botswana. Given that there are currently few cases of COVID-19 diagnosed in both countries, the project will document how the virus spreads within susceptible populations. The development of this proposal is highly collaborative and interdisciplinary, with investigators from Namibia and Botswana working closely with colleagues in Europe. We will also work with an NGO in Namibia, Health Poverty Action, to support rapid implementation.

The project includes two studies that will be conducted sequentially. The first study will follow the WHO protocol for household transmission investigations in the context of COVID-19. It will explore transmission frequency and describe the clinical spectrum of disease. Samples collected will also serve as basis for COVID-19 molecular epidemiology and host immunological response. The second study will evaluate the presentation, diagnosis and clinical characteristics of individuals presenting to sentinel health facilities in both countries. The project will have a strong laboratory strengthening component which will enhance COVID-19 laboratory and research capacity. This will include the development of skills and knowledge for diagnostic testing and COVID-19 sequencing and will build scientific and research capacity.

The findings from this project will provide robust data to assist in guiding national responses to COVID-19 in both countries as well as assisting with our understanding of the pathogenesis of the virus in the context of TB and HIV, in turn providing vital information on how to deliver clinical care and how to design therapeutics and vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Household contact study: all household members of Covid-19 index cases in selected areas
* Healthcare facility study: all attendees of selected primary healthcare facilities

Exclusion Criteria:

* Household contact study: non-household members of Covid-19 index cases in selected areas; individuals not giving consent
* Healthcare facility study: individuals not giving consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Household contact study: household members of Covid-19 index cases in one urban and one rural region of Namibia and Botswana, respectively.
  Healthcare facility study: facility attendees at one urban and one rural primary healthcare facility in Namibian and Botswana, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Covid-19 active infection in households | 6 months
  To determine Covid-19 active infection amongst household members of Covid-19 index cases
Covid-19 active infection in healthcare facilities | 6 months
  To determine Covid-19 active infection amongst healthcare facility attendees

SECONDARY OUTCOMES:
TB infection and disease in households | 6 months
  To determine TB infection and disease amongst household members of Covid-19 index cases
TB infection and disease in healthcare facilities | 6 months
  To determine TB infection and disease amongst healthcare facility attendees
HIV seropositivity in households | 6 months
  To determine HIV seropositivity amongst household members of Covid-19 index cases
HIV seropositivity in healthcare facilities | 6 months
  To determine HIV seropositivity amongst healthcare facility attendees

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Niemann, PhD, Principal Investigator — Research Center Borstel
Locations (1):
- University of Namibia, Windhoek, Namibia

IPD SHARING:
Plan to Share IPD: Undecided